CLINICAL TRIAL: NCT02860585
Title: Evaluation of Survival in Patients With Metastatic Breast Cancer Receiving High-dose Chemotherapy With Autologous Haematopoietic Stem Cell Transplantation
Acronym: BREAST-HDCT
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BREAST-HDCT-IPC 2014-001
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2016-08

CONDITIONS: Breast Neoplasms
Keywords: Metastatic breast cancer; high-dose chemotherapy; autologous haematopoietic progenitor cell transplantation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study was to evaluate the outcome of patients affected with different subtypes of metastatic breast cancer following treatment with high-dose chemotherapy and autologous haematopoietic progenitor cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Metastatic breast Cancer
* Treatment with high-dose chemotherapy and autologous haematopoietic progenitor cell transplantation between 2003 and 2012

Exclusion Criteria:

* Lack of follow-up data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients treated for Metastatic breast Cancer with high-dose chemotherapy and autologous haematopoietic progenitor cell transplantation at the Institut Paoli-Calmettesbetween 2003 and 2012
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival according to Immunohistochemical subtypes . | 8 years

SECONDARY OUTCOMES:
Progression free Survival according to Immunohistochemical subtypes . | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Chabannon, MD,PhD, Study Director — Institut Paoli-Calmettes; Anthony Gonçalves, MD,PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France